CLINICAL TRIAL: NCT00683228
Title: Effect of Using a Structured Tobacco Cessation Education Program in Resident Training on Reducing Secondhand Smoke Exposure in Children
Brief Title: Effect of Using a Structured Tobacco Cessation Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Donna Bacchi, Principal Investigator, State University of New York - Upstate Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5538
Record Dates: First submitted 2008-05-20; First posted 2008-05-23 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Secondhand Smoke Exposure
Keywords: Second hand Smoke
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Counseling (Other): some caregivers will be provided counseling related to the hazards of secondhand smoke exposure
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Counseling — Consecutive newborns exposed to secondhand smoke will be recruited into the study and randomized to have parents receive or not receive specific counselling on harmful effects of SHS exposure. Urine cotinine will be measured at several points during the study for each group

SUMMARY:
This is a pilot study that aims to

1. Evaluate the effectiveness of using a structured tobacco cessation education program, CEASE (Clinical effort against second hand smoke exposure), NY, delivered by pediatric residents in the outpatient continuity clinic of the pediatric residency program in reducing the exposure of infants to second hand smoke.
2. Evaluate the efficacy of using a second hand smoke exposure biomarker, Urine cotinine level measurement and feedback as an adjunct to counseling.

DETAILED DESCRIPTION:
The WHO estimates that half the children in the world are exposed to secondhand smoke. Despite recent smoke free legislation across the country, an estimated 22 percent of children are still exposed in their home environments. These children have increased rates of lower respiratory illnesses, middle ear effusion, asthma, reduced lung function and SIDS. This study aims to evaluate the effectiveness of using a structured tobacco cessation education program, CEASE (Clinical Effort against Secondhand Smoke Exposure), delivered by pediatric residents in the outpatient continuity clinic of a pediatric residency program in reducing the exposure of infants to secondhand smoke. It will also evaluate the efficacy of using a secondhand smoke biomarker, urine cotinine level measurement and feedback as an adjunct to counseling.

Residents(and faculty) whose continuity clinic will be doing the intervention will be receiving tailored training on CEASE NY. The control continuity residents and faculty will receive no additional training. Pre and Post test questionnaires will be administered to all residents of both continuity clinics to test effectiveness of the teaching intervention and use of cotinine level on knowledge and practice. Consecutive newborns with a history of smoking in their home will be recruited into the study ( 22 in each group) when they first establish care ( between days 3 and 15), using a screening question on the nurses portion of the well child form. The study coordinator will obtain consent for participation from those screening positive for smoking in the home. Once consent is obtained the newborns will be randomly assigned to either intervention or control group by the study coordinator. The intervention group will be assigned to a CEASE trained resident for follow-up continuity care. The controls will be assigned to a non- CEASE trained resident for follow-up care. The study coordinator will log the date, agreement/non-agreement to participate, and who the caregiver is (parent vs. other) and to what group they have been assigned, giving them a unique study number. To account for the possibility of dropout, we will recruit 22 infants into each group. Baseline urine samples will be obtained for both groups. The intervention group will receive specific CEASE materials (see attached) and counseling at 2, 4, 6, month well child visits and urine for cotinine will be obtained at 4 and 9 months. Intervention parents will be given feedback on the urine cotinine levels at the next well child visit. The control group will receive no intervention at 2, 4, 6 months. A urine cotinine level will be obtained and a follow-up questionnaire will be given at the 9 month visit to both group parents evaluating their readiness to quit/cut down smoking and their subjective perception of the efficacy of resident counseling.

Baseline urine samples will be obtained for both groups. The intervention group will receive specific CEASE materials (see attached) and counseling at 2, 4, 6, month well child visits and urine for cotinine will be obtained at 4 and 9 months. Intervention parents will be given feedback on the urine cotinine levels at the next well child visit. Control Group will receive no intervention at 2, 4, 6 months. A urine cotinine level will be obtained and a follow-up questionnaire will be given at the 9 month visit to both group parents evaluating their readiness to quit/cut down smoking and their subjective perception of the efficacy of resident counseling. All children will receive a small age-appropriate toy at the 12 month well child check as a thank you for participating in the study

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants up to 15 days of age

Exclusion Criteria:

* Non English speaking family and infants with significant medical problems at birth needing NICU stay
* foster children and wards of state

Ages: 1 Day to 15 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of using a structured tobacco cessation education program, CEASE,delivered by pediatric residents in the outpatient continuity clinic of the pediatric residency program in reducing the exposure of infants to second hand smoke. | Begining of study and at completion of study

SECONDARY OUTCOMES:
Evaluate the efficacy of using a second hand smoke exposure biomarker, Urine cotinine level measurement and feedback as an adjunct to counseling | first visit, 4 month visit, 9 month visit

CONTACTS AND LOCATIONS:
Overall Officials: Donna Bacchi, Md, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States